CLINICAL TRIAL: NCT03612011
Title: Evaluation of the Restorative Efficacy of the Cosmetic Product "Onco-Repair" vs. Placebo on Grade 2 Hand Foot Syndrome Induced by Targeted Therapies or Conventional Chemotherapy. Randomized, Multicentre, Double Blind, Controlled Study Versus Placebo.
Brief Title: Efficacy of the Cosmetic Product "Onco-Repair" on Grade 2 Hand Foot Syndrome
Acronym: OCRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Quanta Medical (Industry)
Collaborators: NAOS Institute of Life Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAOS_ONCOREPAIR_PP_17_2851
Record Dates: First submitted 2018-07-12; First posted 2018-08-02 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Grade 2 Hand-foot Syndrom
Keywords: Hand Foot Syndrome Grade 2; Common Terminology Criteria for Adverse Events (CTCAE); Oncology; Repair Cream; Cutaneous events; Palmar-plantar erythrodysesthesia syndrome; Targeted Therapies or Conventional Chemotherapy
MeSH Terms: conditions — Neoplasms; Hand-Foot Syndrome

STUDY DESIGN:
Intervention Model Description: Phase III multicenter, double blind, superiority, prospective, randomised controlled study Subjects will be randomized to receive either cosmetic product "Onco-Repair" or placebo in a 1:1 ratio
Who Masked: Participant, Investigator
Masking Description: Cosmetic product "Onco-Repair" and placebo will be filled in the tubes with same appearance and smell. The tubes will be marked anonymusioly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onco-Repair (Experimental): Onco-Repair tube of 150 ml
  Interventions: Other: Onco-Repair/ Placebo
- Placebo (Placebo Comparator): Placebo tube of 150 ml
  Interventions: Other: Onco-Repair/ Placebo

INTERVENTIONS:
Other: Onco-Repair/ Placebo — Cream must be applied twice a day, in the morning and evening, on the hands and feet (palmo-plantar areas and interdigital spaces included) previously cleaned with Atoderm Intensive Foaming Gel, chosen as a standardized hygiene product.

SUMMARY:
The aim of the study is to assess the restorative efficacy of the cosmetic product "Onco-Repair" vs placebo of the most affected palmer face in subject with grade 2 HFS induced by targeted therapies or conventional chemotherapy.

DETAILED DESCRIPTION:
HFS, also known as Palmar-Plantar Erythrodysethesia, is a common adverse event observed in subjects under anti-tumor therapy with conventional chemotherapy or targeted thérapies. The initial symptoms are dysesthesia and tingling in the palms, fingers and soles of feet and erythema, which may progress to burning pain with dryness, cracking, desquamation, ulceration and oedema. Sensory impairment, paresthesia and pruritus have also been reported. Palms of the hands are more frequently affected than soles of the feet, and might even be the only area affected in some subjects.

Although HFS is rarely life-threatening, the skin changes are often painful and debilitating and can impair with the general activities of daily living and quality of life. No standard prevention for HFS has not been established yet.

Onco-Repair is a nourishing and repairing cream specially formulated to treat grade 2 HFS which demonstrate skin tolerance, hypoallergenicity and efficacy through several preclinical and clinical studies on healthy subjects.

Therefore, a randomized, double-blind, placebo-controlled study will be conducted to evaluate efficacy and safety of topical cream 'Onco-Repair' on HFS.

ELIGIBILITY:
Inclusion Criteria:

* Who suffers from grade 2 HFS
* Subject under anti-tumor treatment known to cause this toxicity: targeted therapies or conventional chemotherapy: 5-Fluorouracile, Aflibercept, Axitinib, Bévacizumab, Capécitabine, Cediranib, Cytarabine, Dabrafenib, Docétaxel, Doxorubicine, Epirubicine, Pazopanib, Sorafenib, Sunitinib, Trastuzumab, Regorafenib, Vemurafenib and any other anti-tumor treatment that may lead to this toxicity
* Subject 18 years old and more
* Subject having been informed, having signed a free, informed and written consent
* Woman of childbearing age using contraception deemed effective

Non-Inclusion Criteria:

* Pregnant or lactating women
* Subject having a history of allergic contact dermatitis or irritation to any of the components of the investigational products
* Subjects with another skin pathology that may interfere with the evaluation of a HFS (at the investigator's discretion)
* Subject under anti-inflammatory treatment
* Subject participating in another clinical study during the duration of the study, except in a study assessing one of the molecules listed in the section above
* Subject who has already been treated for Grade 2 HFS or under other local treatment or cosmetic product
* Subject refusing to interrupt the application of his/her usual care
* Subject having a strongly altered general condition and / or non-autonomous subject (Karnofsky index <50%)
* Subject in linguistic or psychic impossibility to understand and sign informed consent or in the impossibility of submitting to the medical follow-up of the study
* Subject deprived of liberty by administrative or judicial decision, or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Overall success | 28 days
  A subject is considered to have attained success if he achieves at least one grade improvement in HFS for the most affected palmer face according to the National Cancer Institute CTCATE V5.0 at any time during study period (28 days).
  The subjects will be defined in success or failure according to the following rules:
  Success: switch from grade 2 to grade 1 or grade 0 Failure: switch from grade 2 to grade 3 If subjects remain at grade 2 at the end of the study, they will be classified as either success or failure according to the evolution of clinical signs and / or quality of life assessed using the Dermatological Life Quality Index (DLQI) scale from D0 to D28.

SECONDARY OUTCOMES:
Time to onset of grade 1 or 0 will be assessed using time (in days) from study commencement (inclusion, D0) to first occurrence of grade 1 or lower HFS according to the CTCAEV5.0 | 28 days
  Time to onset of grade 1 or 0 will be assessed using time (in days) from study
Clinical parameters such as lesion color | Day 0 (inclusion) , Day 7 and Day 28
  Clinical parameters such as lesion color will be assessed
  * On e-CRF at D0, D7 and D28
  * from D0 to D28 using a standardized diary completed by subjects
Clinical parameters such as presence of blisters | Day 0 (inclusion) , Day 7 and Day 28
  Clinical parameters such as presence of blisters will be assessed
  * On e-CRF at D0, D7 and D28
  * from D0 to D28 using a standardized diary completed by subjects
Clinical parameters such as fissures/cracks | Day 0 (inclusion) , Day 7 and Day 28
  Clinical parameters such as fissures/cracks will be assessed
  * On e-CRF at D0, D7 and D28
  * from D0 to D28 using a standardized diary completed by subjects
Assessment of quality of life from D0 to D28 using Dermatology Life Quality Index scale | 28 days
  Quality of life will be assessed from D0 to D28 using Dermatology Life Quality Index scale. It is a simple 10-question validated questionnaire that has been used in over 40 different skin conditions in over 80 countries and is available in over 90 languages.
  Meaning of Dermatology Life Quality Index scale Scores:
  0 to 1 = no effect at all on patient's life 2 to 5 = small effect on patient's life 6 to 10 = moderate effect on patient's life 11 to 20 = very large effect on patient's life 21 to 30 = extremely large effect on patient's life
Assessment of symptoms | Day 0 (inclusion) , Day 7 and Day 28
  Such as intensity of lesions, feeling of subjects, etc will be assessed: on e-CRF at D0, D7 and D28, from D0 to D28 using a standardized diary completed by subjects
Assessment of pain score and prurit at D0, D7 and D28 using a 100 Visual Analogue Scale [Visual analogue scale, 0 (no pain, no prurit) and 100 (worst possible pain or prurit)] | Day 0 (inclusion) , Day 7 and Day 28
  Pain score and prurit will be assessed at D0, D7 and D28 using a 100 Visual Analogue Scale [Visual analogue scale , 0 (no pain, no prurit) and 100 (worst possible pain or prurit)]
Assessment of the repair quality of skin | Day 0 (inclusion) , Day 7 and Day 28
  The repair quality of skin will be assessed from D0, D7 and D28 using a standardized diary completed by subjects.
Cosmetic parameters such as nourishing power of the cream will be assessed at D28 using a standardized diary | 28 days
  Nourishing power will be assessed at D28 using a standardized diary completed by subjects.
Cosmetic parameters such as soothing power of the cream will be assessed at D28 using a standardized diary | 28 days
  Soothing power will be assessed at D28 using a standardized diary completed by subjects.
Cosmetic parameters such as penetration power of the cream will be assessed at D28 using a standardized diary | 28 days
  Penetration power will be assessed at D28 using a standardized diary completed by subjects.
Assessment of compliance | 28 days
  The compliance will be assessed at the end of the study: subject will be considered to be compliant if he/she applied at least the theoretical consumption of 60% of the product.
The overall tolerance will be assessed by the investigator (Subject interrogation). This evaluation will be carried out during visits using the following rating: 1 = Very good tolerance 2 = Good tolerance 3 = Middle tolerance 4 = Poor tolerance | 28 days
  1. = Very good tolerance: no functional signs of discomfort and no objective signs during examination
  2. = Good tolerance: some functional signs of minimal and transient discomfort that did not interrupt the applications and no objective signs during examination
  3. = Middle tolerance: functional signs of discomfort, net or persistent, or objective signs during examination that did not interrupt the applications of the investigationalproduct
  4. = Poor tolerance: functional and / or objectives signs leading to discontinuation of the use of the investigational product
Safety will be will be evaluated in terms of: - the number of subjects presenting during the study period at least : One AE/ One SAE - the total number of AEs during the study period - the total number of SAEs during the study period | 28 days
  Safety will be assessed on the basis of adverse event (AE) reports

CONTACTS AND LOCATIONS:
Locations (1):
- Quanta Medical, Rueil-Malmaison, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lipworth AD, Robert C, Zhu AX. Hand-foot syndrome (hand-foot skin reaction, palmar-plantar erythrodysesthesia): focus on sorafenib and sunitinib. Oncology. 2009;77(5):257-71. doi: 10.1159/000258880. Epub 2009 Nov 16. PMID 19923864
- [Background] Zhang RX, Wu XJ, Lu SX, Pan ZZ, Wan DS, Chen G. The effect of COX-2 inhibitor on capecitabine-induced hand-foot syndrome in patients with stage II/III colorectal cancer: a phase II randomized prospective study. J Cancer Res Clin Oncol. 2011 Jun;137(6):953-7. doi: 10.1007/s00432-010-0958-9. Epub 2010 Nov 27. PMID 21113620